CLINICAL TRIAL: NCT00451828
Title: Cholesterol and Pharmacogenetic Study
Acronym: CAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); San Francisco General Hospital (Other); University of California, Los Angeles (Other); Cedars-Sinai Medical Center (Other); University of Washington (Other); Duke University (Other)
Responsible Party: Ronald M. Krauss, MD, Children's Hospital Oakland Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MM2277
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Hyperlipidemia; Hypercholesterolemia; Coronary Heart Disease; Cardiovascular Disease
Keywords: Statins; Cholesterol; Pharmacogenetics
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia; Coronary Disease; Cardiovascular Diseases | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Simvastatin — 40mg/day

SUMMARY:
The overall objective of the CAP study was to determine genetic influences on efficacy of simvastatin treatment with regard to LDL cholesterol reduction and changes in other markers of cardiovascular disease risk.

DETAILED DESCRIPTION:
Despite widespread use of statin therapy for reducing risk of cardiovascular disease risk, there is considerable inter-individual variation in statin efficacy, and it would be desirable to identify markers that would be predictive of the magnitude of beneficial response. The effect of statin most strongly associated with improved clinical outcomes is reduction in LDL cholesterol. The CAP study was a six week non-randomized, open label study of simvastatin 40 mg/day in a group of 335 African-American and 609 Caucasian volunteer subjects. Measurements of plasma lipids and lipoproteins, as well as other markers of cardiovascular disease risk, were obtained at the screening and entry visits, and after four and six weeks of simvastatin treatment. Both baseline measurements and changes in response to simvastatin therapy are being used to test for associations with genetic polymorphisms. Significant findings are being replicated in other study cohorts.

ELIGIBILITY:
Inclusion Criteria:

* at least 30 years of age
* Total Cholesterol between 160 to 400 mg/dl
* > 3 grandparents of African-American descent or > 3 grandparents of Caucasian descent
* serum triglycerides < 400 mg/dl
* fasting glucose < 126 mg/dl

Exclusion Criteria:

* Use of lipid-lowering medication
* Use of over-the-counter products containing sterol or stanol esters or fish oil
* Recent or planned change in dietary intake or weight change of more than 4.5 kg
* Use of corticosteroids, immunosuppressive drugs or drugs affecting the CYP3A4 system
* Known liver disease or elevated transaminase levels
* Elevated creatine phosphokinase levels > 10 times upper limits of normal
* Uncontrolled blood pressure, or diabetes mellitus
* Abnormal renal or thyroid function
* Current alcohol or drug abuse
* Major illness in the preceding three months
* Pregnancy
* Know intolerance to statins
* Racial ancestry other than African-American or Caucasian

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2002-03; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol | -2, 0, 4, 6 weeks
LDL Cholesterol | -2, 0, 4, 6 weeks
HDL Cholesterol | -2, 0, 4, 6 weeks
Triglycerides | -2, 0, 4, 6 weeks
C-reactive protein | -2, 0, 4, 6 weeks

SECONDARY OUTCOMES:
Total Cholesterol/HDL Cholesterol | -2, 0, 4, 6 weeks
Apolipoprotein B | -2, 0, 4, 6 weeks
Apolipoprotein AI | -2, 0, 4, 6 weeks
Apolipoprotein CIII | -2, 0, 4, 6 weeks
LDL Peak Particle size | -2, 0, 4, 6 weeks
LDL Subfractions | -2, 0, 4, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Simon JA, Lin F, Hulley SB, Blanche PJ, Waters D, Shiboski S, Rotter JI, Nickerson DA, Yang H, Saad M, Krauss RM. Phenotypic predictors of response to simvastatin therapy among African-Americans and Caucasians: the Cholesterol and Pharmacogenetics (CAP) Study. Am J Cardiol. 2006 Mar 15;97(6):843-50. doi: 10.1016/j.amjcard.2005.09.134. Epub 2006 Jan 27. PMID 16516587
- [Derived] Theusch E, Ting FY, Qin Y, Stevens K, Naidoo D, King SM, Yang NV, Orr J, Han BY, Cyster JG, Chen YI, Rotter JI, Krauss RM, Medina MW. Participant-derived cell line transcriptomic analyses and mouse studies reveal a role for ZNF335 in plasma cholesterol statin response. Genome Med. 2024 Jul 26;16(1):93. doi: 10.1186/s13073-024-01366-9. PMID 39061094
- [Derived] Theusch E, Ting FY, Qin Y, Stevens K, Naidoo D, King SM, Yang N, Orr J, Han BY, Cyster JG, Chen YI, Rotter JI, Krauss RM, Medina MW. Participant-derived cell line transcriptomic analyses and mouse studies reveal a role for ZNF335 in plasma cholesterol statin response. bioRxiv [Preprint]. 2023 Jun 15:2023.06.14.544860. doi: 10.1101/2023.06.14.544860. PMID 37397985
- [Derived] Trupp M, Zhu H, Wikoff WR, Baillie RA, Zeng ZB, Karp PD, Fiehn O, Krauss RM, Kaddurah-Daouk R. Metabolomics reveals amino acids contribute to variation in response to simvastatin treatment. PLoS One. 2012;7(7):e38386. doi: 10.1371/journal.pone.0038386. Epub 2012 Jul 9. PMID 22808006
- [Derived] Mangravite LM, Medina MW, Cui J, Pressman S, Smith JD, Rieder MJ, Guo X, Nickerson DA, Rotter JI, Krauss RM. Combined influence of LDLR and HMGCR sequence variation on lipid-lowering response to simvastatin. Arterioscler Thromb Vasc Biol. 2010 Jul;30(7):1485-92. doi: 10.1161/ATVBAHA.110.203273. Epub 2010 Apr 22. PMID 20413733
- [Derived] Barber MJ, Mangravite LM, Hyde CL, Chasman DI, Smith JD, McCarty CA, Li X, Wilke RA, Rieder MJ, Williams PT, Ridker PM, Chatterjee A, Rotter JI, Nickerson DA, Stephens M, Krauss RM. Genome-wide association of lipid-lowering response to statins in combined study populations. PLoS One. 2010 Mar 22;5(3):e9763. doi: 10.1371/journal.pone.0009763. PMID 20339536
- [Derived] Medina MW, Gao F, Ruan W, Rotter JI, Krauss RM. Alternative splicing of 3-hydroxy-3-methylglutaryl coenzyme A reductase is associated with plasma low-density lipoprotein cholesterol response to simvastatin. Circulation. 2008 Jul 22;118(4):355-62. doi: 10.1161/CIRCULATIONAHA.108.773267. Epub 2008 Jun 16. PMID 18559695
- [Derived] Krauss RM, Mangravite LM, Smith JD, Medina MW, Wang D, Guo X, Rieder MJ, Simon JA, Hulley SB, Waters D, Saad M, Williams PT, Taylor KD, Yang H, Nickerson DA, Rotter JI. Variation in the 3-hydroxyl-3-methylglutaryl coenzyme a reductase gene is associated with racial differences in low-density lipoprotein cholesterol response to simvastatin treatment. Circulation. 2008 Mar 25;117(12):1537-44. doi: 10.1161/CIRCULATIONAHA.107.708388. Epub 2008 Mar 10. PMID 18332269